CLINICAL TRIAL: NCT03176927
Title: Biomagnetic Characterization of Gastric Dysrhythmias III
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Alan Bradshaw, Research Assistant Professor of Surgery, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB# 121501; R01DK058697 (NIH)
Record Dates: First submitted 2017-04-05; First posted 2017-06-06 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2023-10

CONDITIONS: Diabetics Without Symptoms of Gastroparesis; Diabetic Gastroparesis; Idiopathic Gastroparesis; Total or Partial Gastrectomy; Chronic Nausea; Functional Dyspepsia
Keywords: magnetogastrogram; gastroparesis; electrogastrogram; gastric slow wave
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Gastroparesis (Experimental): magnetogastrogram
  Diabetes with and without gastroparesis ; Idiopathic gastroparesis
  Interventions: Diagnostic Test: magnetogastrogram
- Gastrectomy (Experimental): magnetogastrogram
  Total or partial gastrectomy group
  Interventions: Diagnostic Test: magnetogastrogram
- Functional dyspepsia (Experimental): magnetogastrogram
  Children with functional dyspepsia
  Interventions: Diagnostic Test: magnetogastrogram
- Chronic nausea (Experimental): magnetogastrogram
  Children with chronic nausea
  Interventions: Diagnostic Test: magnetogastrogram
- Control participants (Experimental): magnetogastrogram
  Group without any gastrointestinal diseases.
  Interventions: Diagnostic Test: magnetogastrogram

INTERVENTIONS:
Diagnostic Test: magnetogastrogram

SUMMARY:
There is a tremendous clinical need for a noninvasive technique that can assess gastric electrical activity and would be repeatable without any exposure to radiation. Investigators developed a new technique allowing to use noninvasive methods to assess bioelectrical activity in the gastrointestinal system. This has enabled to characterize the normal and pathologic physiology of the stomach through the use of noninvasive magnetogastrogram (MGG) records. Primary hypothesis for this proposal is that analysis of gastric slow wave uncoupling and propagation in multichannel MGG discriminates between normal and pathological gastric electrical activity. Eventually, investigators envision this research leading to new insights for gastrointestinal conditions such as gastroparesis, functional dyspepsia and chronic idiopathic nausea that would inform clinical management of these debilitating diseases.

DETAILED DESCRIPTION:
5/23/25. Study record updated to reflect Early Phase 1/Phase 0 trial. The main aim of the study was to evaluate MGG as a device for classification of functional gastric disorders.

Studies have demonstrated that the magnetogastrogram (MGG) records the same gastric slow wave activity that detect with serosal and mucosal electrodes. The upgraded magnetometer will improve the spatial resolution resulting in increased sensitivity for detecting and characterizing both abnormal frequency dynamics and abnormal spatiotemporal patterns. The spatiotemporal data collected with multichannel Superconducting QUantum Interference Device (SQUID) biomagnetometer has allowed , for the first time, to characterize propagation of the gastric slow wave noninvasively. In addition to frequency dynamic changes, which are the only reliable parameters from cutaneous electrogastrogram (EGG), and which still do not necessarily correlate well with disease, the MGG reflects normal and abnormal gastric slow wave activity. Furthermore, for the first time, investigators have demonstrated that propagation characteristics determined magnetically distinguish normal subjects from patients with gastroparesis. Also for the first time, investigators have been able to detect the gradient in gastric propagation velocity noninvasively in animal subjects. However, investigators still have unresolved questions about how MGG propagation rhythm and pattern disturbances may specify functional disorders.

ELIGIBILITY:
Inclusion Criteria:

* Participants between ages 12-80
* Diabetic patients with gastroparesis, diabetic patients without gastroparesis and who are willing to have a gastric emptying test if they have not had one in the last 6 months and an IV inserted.
* Patients with idiopathic gastroparesis
* Total or partial gastrectomy patients
* Children (ages 12-17) with functional dyspepsia
* Children (ages 12-17) with chronic nausea

Exclusion Criteria:

* Those with claustrophobia who cannot lie still under the SQUID for the length of time required.
* Normal participants with known intestinal complications
* Pregnant females (females who are able to have children will be given a pregnancy test).
* Morbid obesity (these patients are presumably unable to lie under the current generation of SQUID devices).
* Patients with a history of cardiac arrhythmias, taking anticoagulants, or greater than 80 years of age will be excluded.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-12; Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Measurement of gastric slow wave activity in normal and diseased smooth muscle of the stomach | 1 day

SECONDARY OUTCOMES:
Measurement of gastric slow wave propagation velocity in gastroparesis patients | 1 day
Measurement of invasive serosal electromyogram before and after partial/total gastrectomy. | day 1 and day 30
Measurement of noninvasive magnetogastrogram before and after partial/total gastrectomy. | day 1 and day 30
Noninvasive measurement of gastric slow wave dysrhythmia in pediatric patients with nausea and functional dyspepsia | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Leonard A Bradshaw, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradshaw LA, Cheng LK, Chung E, Obioha CB, Erickson JC, Gorman BL, Somarajan S, Richards WO. Diabetic gastroparesis alters the biomagnetic signature of the gastric slow wave. Neurogastroenterol Motil. 2016 Jun;28(6):837-48. doi: 10.1111/nmo.12780. Epub 2016 Feb 3. PMID 26839980
- [Background] Bradshaw LA, Kim JH, Somarajan S, Richards WO, Cheng LK. Characterization of Electrophysiological Propagation by Multichannel Sensors. IEEE Trans Biomed Eng. 2016 Aug;63(8):1751-9. doi: 10.1109/TBME.2015.2502065. Epub 2015 Nov 19. PMID 26595907
- [Background] Kim JH, Pullan AJ, Bradshaw LA, Cheng LK. Influence of body parameters on gastric bioelectric and biomagnetic fields in a realistic volume conductor. Physiol Meas. 2012 Apr;33(4):545-56. doi: 10.1088/0967-3334/33/4/545. Epub 2012 Mar 14. PMID 22415019
- [Background] Somarajan S, Cassilly S, Obioha C, Richards WO, Bradshaw LA. Effects of body mass index on gastric slow wave: a magnetogastrographic study. Physiol Meas. 2014 Feb;35(2):205-15. doi: 10.1088/0967-3334/35/2/205. Epub 2014 Jan 7. PMID 24398454
- [Background] Somarajan S, Muszynski ND, Obioha C, Richards WO, Bradshaw LA. Biomagnetic and bioelectric detection of gastric slow wave activity in normal human subjects--a correlation study. Physiol Meas. 2012 Jul;33(7):1171-9. doi: 10.1088/0967-3334/33/7/1171. Epub 2012 Jun 27. PMID 22735166